CLINICAL TRIAL: NCT05579145
Title: Effects of Combined Tracheal Suctioning and Expiratory Pause 5 or 10 Seconds: a Crossover Randomized Clinical Trial
Brief Title: Tracheal Suctioning and Expiratory Pause in Bronchial Hygiene
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 51995621.7.0000.5327
Record Dates: First submitted 2022-09-21; First posted 2022-10-13 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Mechanical Ventilation
Keywords: Bronchial hygiene; Tracheal suctioning; Respiratory therapy; Intensive care unit

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-Second Expiratory Pause (Experimental): Closed system aspiration following by expiratory pause with mechanical ventilator for 5 seconds.
  Interventions: Other: 5-Second Expiratory Pause
- 10-Second Expiratory Pause (Experimental): Closed system aspiration following by expiratory pause with mechanical ventilator for 10 seconds.
  Interventions: Other: 10-Second Expiratory Pause

INTERVENTIONS:
Other: 5-Second Expiratory Pause — Patients on mechanical ventilation for more than 24 hours will be randomized for the first technique to be applied. This technique consists of closed system aspiration and expiratory pause with mechanical ventilator for 5 seconds. After randomization and before the application of the technique, all patients will be positioned in supine position with the headboard elevated at 30 degrees and will be aspirated once with closed aspiration system and with vacuum of -40 cm H2O.
  Arms: 5-Second Expiratory Pause
Other: 10-Second Expiratory Pause — Patients on mechanical ventilation for more than 24 hours will be randomized for the first technique to be applied. This technique consists of closed system aspiration and expiratory pause with mechanical ventilator for 10 seconds. After randomization and before the application of the technique, all patients will be positioned in supine position with the headboard elevated at 30 degrees and will be aspirated once with closed aspiration system and with vacuum of -40 cm H2O.
  Arms: 10-Second Expiratory Pause

SUMMARY:
A randomized crossover clinical trial conducted in an Intensive Care Unit of the Hospital de Clinicas de Porto Alegre (HCPA) to compare the efficacy of the two techniques on the amount of aspirated pulmonary secretion and pulmonary mechanics: aspiration of the closed system following an expiratory pause with mechanical ventilator for 5 seconds (5-Second Expiratory Pause) and aspiration of the closed system following an expiratory pause with mechanical ventilator for 10 seconds (10-Second Expiratory Pause).

DETAILED DESCRIPTION:
After randomization, all patients will be positioned in dorsal decubitus with the head elevated at 30 degrees and will be aspirated once with a closed suction system and with a vacuum of -40cm H2O. Hemodynamic and pulmonary parameters will be collected and recorded. One of the two techniques will be applied, according to randomization, and the outcomes measured. After two hours, hemodynamic and pulmonary parameters will be re-collected, and the second technique will be applied. The outcomes will be measured again.

ELIGIBILITY:
Inclusion Criteria:

* Patients in 24 and 72 hours of mechanical ventilation.
* Patients with closed aspiration system.
* Patients hemodynamically stable (mean arterial blood pressure ≥ 60 mmHg and with dose of Noradrenaline ≤ 1μg/kg/minute).

Exclusion Criteria:

* Undrained pneumothorax and hemothorax.
* Subcutaneous emphysema.
* Patients who refuse to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Weight of secretion aspirated (grams) | Immediately after the application of one of the closed system aspiration techniques.
  The secretion aspirated into the collection flask will be weighed on a precision laboratory scale.

SECONDARY OUTCOMES:
Peripheral arterial oxygen saturation (SpO2) (%) | One minute after the application of the studied technique.
  After the 3-second expiratory pause on the mechanical ventilator, the SpO2 will be visualized on the monitor of the patient, and the value will be noted.
Peak inspiratory pressure (PIP) (cm H2O) | One minute after the application of the studied technique.
  The PIP will be visualized directly at mechanical ventilation monitor, and the value will be noted.
End expiratory pressure (PEEP) (cmH2O) | One minute after the application of the studied technique.
  The PEEP will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Air trapping (AUTO-PEEP) (cmH2O) | One minute after the application of the studied technique.
  The AUTO-PEEP will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Mechanical ventilation circuit pressure (cmH2O) | One minute after the application of the studied technique.
  The mechanical ventilation circuit pressure will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Tidal volume (TV) (ml) | One minute after the application of the studied technique.
  The TV will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Endotracheal tube diameter (ETT) (mm) | One minute after the application of the studied technique.
  The endotracheal tube diameter is directly written in the product package.
Dynamic compliance (Cd) (ml/cmH2O) | One minute after the application of the studied technique.
  The Cd will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Resistance (R) (L/s) | One minute after the application of the studied technique.
  The R will be visualized directly at mechanical ventilation monitor, and the value will be noted.
Drive pressure (cmH2O) | One minute after the application of the studied technique.
  The drive pressure will be calculated by the difference between plateau pressure and positive end-expiratory pressure in the mechanical ventilation, and the value will be noted.
Heart rate (HR) (beats per minute) | One minute after the application of the studied technique.
  After the 3-second expiratory pause on the mechanical ventilator, the HR will be visualized on the monitor of the patient, and the value will be noted.
Respiratory rate (RR) (breaths per minute). | One minute after the application of the studied technique.
  After the 3-second expiratory pause on the mechanical ventilator, the RR will be visualized on the monitor of the patient, and the value will be noted.
Mean arterial pressure (MAP) (mmHg) | One minute after the application of the studied technique.
  After the 3-second expiratory pause on the mechanical ventilator, the MAP will be calculated using the systolic and diastolic blood pressure, and the value will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Luciane FG Martins, Master, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (2):
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Luciane FG Martins, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Background] McCarren B, Alison JA, Herbert RD. Manual vibration increases expiratory flow rate via increased intrapleural pressure in healthy adults: an experimental study. Aust J Physiother. 2006;52(4):267-71. doi: 10.1016/s0004-9514(06)70006-x. PMID 17132121
- [Background] Amato MB, Carvalho CR, Isola A, Vieira S, Rotman V, Moock M, Jose A, Franca S. [Mechanical ventilation in Acute Lung Injury (ALI)/Acute Respiratory Discomfort Syndrome (ARDS)]. J Bras Pneumol. 2007;33 Suppl 2S:S119-27. doi: 10.1590/s1806-37132007000800007. No abstract available. Portuguese. PMID 18026670
- [Background] Bhowmik A, Chahal K, Austin G, Chakravorty I. Improving mucociliary clearance in chronic obstructive pulmonary disease. Respir Med. 2009 Apr;103(4):496-502. doi: 10.1016/j.rmed.2008.10.014. Epub 2008 Dec 16. PMID 19091536
- [Background] Ntoumenopoulos G, Presneill JJ, McElholum M, Cade JF. Chest physiotherapy for the prevention of ventilator-associated pneumonia. Intensive Care Med. 2002 Jul;28(7):850-6. doi: 10.1007/s00134-002-1342-2. Epub 2002 May 24. PMID 12122521
- [Background] Van der Schans CP. Bronchial mucus transport. Respir Care. 2007 Sep;52(9):1150-6; discussion 1156-8. PMID 17716383
- [Background] Sarmento, GJ et al. Fisioterapia em UTI: Avaliação e Procedimentos. Editora Atheneu.Vol 1. São Paulo, 2006. Págs: 353.
- [Background] Ciesla ND. Chest physical therapy for patients in the intensive care unit. Phys Ther. 1996 Jun;76(6):609-25. doi: 10.1093/ptj/76.6.609. PMID 8650276
- [Background] Savian C, Paratz J, Davies A. Comparison of the effectiveness of manual and ventilator hyperinflation at different levels of positive end-expiratory pressure in artificially ventilated and intubated intensive care patients. Heart Lung. 2006 Sep-Oct;35(5):334-41. doi: 10.1016/j.hrtlng.2006.02.003. PMID 16963365
- [Background] Carlon GC, Fox SJ, Ackerman NJ. Evaluation of a closed-tracheal suction system. Crit Care Med. 1987 May;15(5):522-5. doi: 10.1097/00003246-198705000-00015. PMID 3552445
- [Background] Mattar JA, Sproesser AM, Gomes MA. A comparative study of oxygen transport between open and closed methods of tracheal suctioning. Intensive and Critical Care Digest, 1992.
- [Background] Craig KC, Benson MS, Pierson DI. Prevention of arterial oxygen desaturation during closed-airway endotracheal suction: effect of ventilator mode. Resp. Care, v. 29, p. 103-7, 1984
- [Background] Deppe SA, Kelly JW, Thoi LL, Chudy JH, Longfield RN, Ducey JP, Truwit CL, Antopol MR. Incidence of colonization, nosocomial pneumonia, and mortality in critically ill patients using a Trach Care closed-suction system versus an open-suction system: prospective, randomized study. Crit Care Med. 1990 Dec;18(12):1389-93. doi: 10.1097/00003246-199012000-00016. PMID 2245613
- [Background] Ritz R, Scott LR, Coyle MB, Pierson DJ. Contamination of a multiple-use suction catheter in a closed-circuit system compared to contamination of a disposable, single-use suction catheter. Respir Care. 1986 Nov;31(11):1086-91. PMID 10315714
- [Background] Taggart JA, Dorinsky NL, Sheahan JS. Airway pressures during closed system suctioning. Heart Lung. 1988 Sep;17(5):536-42. PMID 3417464
- [Background] Pepe PE, Marini JJ. Occult positive end-expiratory pressure in mechanically ventilated patients with airflow obstruction: the auto-PEEP effect. Am Rev Respir Dis. 1982 Jul;126(1):166-70. doi: 10.1164/arrd.1982.126.1.166. PMID 7046541
- [Background] Sarmento GJV, et al. Fisioterapia Respiratória no Paciente Crítico: Rotinas Clínicas. 3° ed. rev e ampl- Barueri /SP. Editora: Manole, 2010.
- [Background] Lemes DA, Zin WA, Guimaraes FS. Hyperinflation using pressure support ventilation improves secretion clearance and respiratory mechanics in ventilated patients with pulmonary infection: a randomised crossover trial. Aust J Physiother. 2009;55(4):249-54. doi: 10.1016/s0004-9514(09)70004-2. PMID 19929767
- [Background] Naue Wda S, da Silva AC, Guntzel AM, Condessa RL, de Oliveira RP, Rios Vieira SR. Increasing pressure support does not enhance secretion clearance if applied during manual chest wall vibration in intubated patients: a randomised trial. J Physiother. 2011;57(1):21-6. doi: 10.1016/S1836-9553(11)70003-0. PMID 21402326
- [Background] Azeredo CA, Bezerra RM. Manobras de Fisioterapia Respiratória na UTI.Editora SOS Pulmão/Cuca. Rio de Janeiro, 2004. Págs: 139.
- [Background] David CM. Medicina Intensiva. Editora Revinter. Rio de Janeiro, 2004. Págs: 1159.
- [Background] de Fraga Gomes Martins L, da Silva Naue W, Skueresky AS, Bianchi T, Dias AS, Forgiarini LA. Effects of Combined Tracheal Suctioning and Expiratory Pause: A Crossover Randomized Clinical Trial. Indian J Crit Care Med. 2019 Oct;23(10):454-457. doi: 10.5005/jp-journals-10071-23263. PMID 31749553